CLINICAL TRIAL: NCT05088564
Title: Pylorus-preserving Pancreaticoduodenectomy Using a Hemi-double-stapling Technique
Brief Title: Efficacy of Hemi-double-stapling Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Joon Seong Park, Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3-2021-0084
Record Dates: First submitted 2021-08-08; First posted 2021-10-22 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Periampullar Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I (Hand-sewn group) (Experimental): Doudenojejunal anastomosis by hand-swen method
  Interventions: Procedure: Hand-sewn
- II (Stapling group) (Active Comparator): Doudenojejunal anastomosis by hemi-double-stapling method
  Interventions: Procedure: Hemi-double stapling

INTERVENTIONS:
Procedure: Hand-sewn — Doudenojejunal anastomosis by hand-sewn method
  Arms: I (Hand-sewn group)
Procedure: Hemi-double stapling — Doudenojejunal anastomosis by hemi-double-stapling method "EEA25 - Covidien EEA Circular Stapler DST Series 25.0mm x 4.8mm" is used for anastomosis
  Arms: II (Stapling group)

SUMMARY:
Surgical stapler is used in all areas of surgical operation. Surgical stapler has been used in various surgical fields for a long time, so its stability has already been proven. After gastrectomy or colectomy, the hemi-double stapling technique, which is an improved double stapling technique, has been applied as an anastomosis method using a stapler.

In the duodenojejunal anastomosis after PPPD, the hemi-double stapling method can be applied to preserve the pyloric branch of the vagus nerve and the branch of the right gastric artery to ensure sufficient blood supply. Ultimately, it is expected to shorten the anastomosis time as well as reduce the frequency of delayed gastric emptying. In addition, the work of physically expanding the pylorus to insert the circular anastomosis is also thought to reduce gastric emptying delay.

DETAILED DESCRIPTION:
(1) Stapling technique

1. Make purse-string suture on jejunum at the point of duodenojejunostomy
2. Insert Anvil into jejunem
3. Make incision of 3-4 centimeters at anterior side of antrum
4. Long Kelly forceps are inserted into the stomach to dilate the pylorus
5. A 25 mm end-to-end anastomosis (EEA) stapler is inserted into the stomach and passed through the pylorus.
6. The needle of EEA stapler is pierced through the lower part of the stapler line where the duodenum has been resected
7. The EEA stapler is combined with the anvil and anastomosis is performed
8. The incision on the stomach is sutured through a linear stapler
9. Reinforcement suture for stapler line

(2) Postoperative management

* Diet build up as same manner of hand-sewn group (3) Postoperative follow-up
* All postoperative complication, delayed gastric emptying, intraperitoneal abscess, postoperative pancreatic fistula, postpancreatectomy hemorrhage, hospital stay, reoperation, readmission and 2-months mortality.

ELIGIBILITY:
Inclusion Criteria:

1. pylorus-preserving pancreaticoduodenectomy
2. ECOG scale 0-1
3. Age > 19
4. Appropriate organ function as below i.WBC : ≥2500 mm3, ≤14000 mm3 ii.Hemoglobin : ≥9.0 g/dL iii.Platelet : ≥100,000 mm3 iv.Total bilirubin : ≤2.0 mg/dL (except for occlusive jaundice) v.Creatinine : ≤2.0 mg/dL
5. patient who can understand and sign the informed consent

Exclusion Criteria:

1. previous history of gastrectomy
2. ulcerative scar around ampulla of duodenum on endoscopy
3. previous history of upper abdomen surgery (open)
4. Emergency
5. Severe ischemic heart disease
6. Severe hepatic failure by liver cirrhosis or hepatitis
7. Severe respiratory failure that requires oxygene inhalation
8. Chronic renal failure that requires hemodialysis
9. Expecting combine resection of other organ
10. Immunosuppressive therapy
11. Accompanying cancer with potential for adverse events
12. Severe psychologic or neurologic disease
13. drug or alcohol addiction

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2024-04-22 (Estimated); Study Completion 2024-04-22 (Estimated)

PRIMARY OUTCOMES:
Grade of delayed gastric emptying by ISGPS | At postoperative 21 day
  Delayed gastric emptying will be evaluated at postoperative 21 day using International study group of pancreatic surgery (ISGPS) classification. According to ISGPS classification, delayed gastric emptying is divided into three grades from A to C. Grade C means worse than grade A.-->Unit of Measure: Grade A,B,C

SECONDARY OUTCOMES:
hospital stay | At postoperative 21 day
  Duration (days) of hospital stay, which means interval between operation day and discharge day will be checked up to postoperative 2 months. --> Unit of Measure: days

OTHER OUTCOMES:
intraperitoneal abscess | at postoperative 2 months
  Intraperitoneal abscess will be evaluated using 2 point scale (yes or no) at postoperative 2 months.
  * Unit of Measure: Yes, No
Incidence of reoperation/ readmission | At postoperative 21 day
  The incidence of reoperation and readmission will be evaluated using 2 point scale (yes or no) at postoperative 2 months.--> Unit of Measure: Yes, No

CONTACTS AND LOCATIONS:
Overall Officials: Joon Seoung Park, Principal Investigator — GangnamSeverance Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No